CLINICAL TRIAL: NCT03059277
Title: Efficacy of Intravitreal Aflibercept Injection (IAI) Administered in a Treat and Extend Fashion in Patients With Center Involved Diabetic Macular Edema (DME) Previously Managed With 0.3 mg Intravitreal Ranibizumab
Brief Title: Intravitreal Alfibercept for Center Involved DME Previously Managed With Intravitreal Ranibizumab
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Site investigator decided to not move forward with study.
Sponsor: Southeast Clinical Research Associates, LLC (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-DME-1432
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Diabetes; reduced treatment frequency
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravitreal Aflibercept (Experimental): Intravitreal Aflibercept Injection (IAI)
  Interventions: Drug: Intravitreal Aflibercept

INTERVENTIONS:
Drug: Intravitreal Aflibercept — Intravitreal Aflibercept 2mg

SUMMARY:
The purpose of this study is to determine the efficacy of intravitreal aflibercept injections administered in a treat and extend fashion in eyes that have persistent center involved diabetic macular edema following at least 4 intravitreal injections of 0.3 mg ranibizumab over 24 weeks.

DETAILED DESCRIPTION:
This is a phase 4 prospective, nonrandomized, open label, interventional clinical trial to determine the efficacy of intravitreal aflibercept (IAI) administered in a treat and extend fashion in eyes that have persistent centered involved diabetic macular edema despite at least 4 intravitreal injections of ranibizumab 0.3mg over 24 weeks prior to enrollment. Patients will receive intravitreal injections of aflibercept (2mg/0.05cc) at baseline and monthly until an eye has reached stability defined as: < 10% change in the Spectral Domain Optical Coherence Tomography (SD OCT) central retinal thickness (CRT) reading from the previous 2 visits (can include baseline) and less than a 5 letter decrease in Best Corrected Visual Acuity (BCVA) from best BCVA from prior visits. Once an eye has reached stability criteria, a treat and extend protocol will be used and treatment will be rendered on every visit. The duration between treatments will be extended by 2 weeks from the last visit if SD OCT extension criteria are met: < 10% change in CRT over 2 consecutive visits and < 5 letter decrease in BCVA from baseline

If at any return visit subretinal and/or intraretinal fluid recurs that causes the CRT to increase by > 10 % from its lowest level in the previous 2 consecutive visits, or CRT increases by < 10% due to subretinal and/or intraretinal fluid but is associated with a decrease of BCVA of > 5 letters from baseline then the eye will receive IAI and the treatment interval will be decreased by 1 week. If the eye has not improved or worsened for at least 2 consecutive visits and the SD OCT central subfield thickness is ≥ 300 microns or visual acuity is worse than 20/20, the following will be done:

Prior to the 24-week visit, an injection will be given. At and after the 24-week visit, an injection will be given and modified grid laser can be given at the discretion of the investigator within 7 days of IAI based on rescue criteria

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years with type 1 or type 2 diabetes
* Best Corrected Visual Acuity (by ETDRS) letter score in study eye ≤ 85 and ≥24 (approximate Snellen equivalent 20/20 to 20/320)
* Central retinal thickness on SD OCT at baseline visit of > 300 microns using Heidelberg Spectralis with definite evidence of intraretinal or subretinal fluid due to diabetic retinopathy in the CSF.
* Patients must have received at least four intravitreal ranibizumab 0.3 mg injections within 24 weeks prior to screening and failed to have had complete resolution of intraretinal or subretinal fluid on SD OCT and a CRT > 300 microns using Heidelberg Spectralis

Exclusion Criteria:

* Laser photocoagulation (panretinal or macular) in the study within 90 days of baseline
* Active high risk proliferative diabetic retinopathy (PDR)
* History of intravitreal corticosteroids within 4 months of baseline
* History of intravitreal bevacizumab within 24 weeks of baseline
* History of idiopathic or autoimmune uveitis in the study eye
* Cataract surgery in the study eye within 90 days of baseline
* Any intraocular surgery within 90 days of baseline
* Vitreomacular traction or epiretinal membrane in the study eye that is thought to affect vision
* Evidence of active infection in either eye
* Uncontrolled glaucoma in the study eye defined as a pressure of > 25 mmHg on maximal medical therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Central Subfield Thickness (CST) | 52 weeks
  Percentage of patients who experience a > 10% decrease in mean Central Subfield Thickness (CST) from baseline or whose CST < 300 microns at 52 weeks.

SECONDARY OUTCOMES:
Mean Change in Visual Acuity | 52 weeks
  Mean change in Best Corrected Visual Acuity
Change in Central Subfield Thickness (CST) | 52 weeks
  Mean change in CST on SD OCT compared to baseline
Number of Intravitreal Injections | 52 Weeks
  Mean number of injections from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrew N Antoszyk, MD, Principal Investigator — Charlotte Eye Ear Nose and Throat Assciates, PA
Locations (2):
- United States (2):
  - Charlotte Eye Ear Nose and Throat Associates, PA, Charlotte, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates, PA, Statesville, North Carolina

IPD SHARING:
Plan to Share IPD: No
Site will not be sharing IPD.